CLINICAL TRIAL: NCT04509531
Title: Development of Resilience Against Cyberbullying Victimization
Brief Title: Building Resilience in Cyberbullying Victims
Acronym: Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Deusto (Other)
Collaborators: Fundación Alicia Koplowitz (Unknown)
Responsible Party: Principal Investigator, Esther Calvete, Principal Investigator, Deusto Stress Research Team, University of Deusto, University of Deusto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019-0000222
Record Dates: First submitted 2020-07-30; First posted 2020-08-12 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Cyberbullying; Depression; Non Suicidal Self Injury; Social Anxiety; Eating Disorders
Keywords: Adolescence; Prevention; Cyberbullying; Depression; Non Suicidal Self Injury; Social Anxiety; Eating Disorders
MeSH Terms: conditions — Cyberbullying; Depression; Self-Injurious Behavior; Feeding and Eating Disorders | interventions — Inosine Triphosphate

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio blocked by gender to one of two groups: experimental condition (SA, ITP and resilience condition) versus control condition (anti-grooming/sexting condition) in parallel for the duration of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Allocation will be concealed to the participants, researchers -who will be in class the assessment days if possible depending on the Covid-19 scenario- and teachers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: SA, ITP and Resilience (Experimental): 1 hour Wise intervention (based on SA, ITP and resilience) consisting on several tasks to be completed online individually.
  Interventions: Behavioral: Wise Intervention (SA, ITP and resilience)
- Standard preventive intervention (Other): 1 hour educational intervention (about internet risks such as sexting and grooming) consisting on several tasks to be completed online individually.
  Interventions: Behavioral: Standard preventive intervention

INTERVENTIONS:
Behavioral: Wise Intervention (SA, ITP and resilience) — The intervention will be based on four general types of change strategies: (1) scientific knowledge, (2) generation of new meanings, (3) commitment through action, and (4) active reflection. This will include activities such as reading scientific information about social behavior and its role in people's well-being and mental health, the meaning of online victimization experiences and ways to react to them, experiences of other young people of their age, and self-persuasion exercises that involve an active commitment to change. Furthermore, it provides a number of strategies to manage everyday conflicts among adolescents. This intervention teaches them new ways to manage these difficulties through different actions (relaxation, distraction, sports, etc.). Finally, they are asked to plan the strategies they will use in the future in the face of some difficulties and to recommend some guidelines for another adolescent who may be going through a similar situation.
  Arms: Experimental: SA, ITP and Resilience
Behavioral: Standard preventive intervention — The control intervention will involve scientific information and education about internet risks such as sexting and grooming.
  Arms: Standard preventive intervention

SUMMARY:
This study evaluates the effectiveness of a wise intervention based on self-affirmation (SA) and Implicit Theories of Personality (ITP) building resilience in victims. Half of the participants will receive the experimental intervention, while the other half will receive a control intervention.

DETAILED DESCRIPTION:
Bullying victimization can harm victims' mental health. Numerous studies have shown that, when an adolescent is a victim of cyberbullying, the risk of developing numerous mental health problems increases. Tackling the problem of cyberbullying victims' worsening mental health involves at least (1) reducing bullying itself, as this would reduce the prevalence of victimization, and (2) building resilience in the victims so that their mental health does not worsen. In recent years, a number of preventive interventions have been developed aimed at reducing cyberbullying but not so much focused on building resilience in the victims. Very recently, interest in scientific social psychology has grown due to a new approach to interventions, which have been called "wise interventions." This approach involves a set of rigorous techniques, based on theory and research, that address specific psychological processes to help people thrive in various life environments. The main objective of this project is to extend the previous findings to the mental health effects of online victimization in adolescents. In this project it will be designed and evaluated the effectiveness of an wise intervention aimed at (1) reducing online bullying, as this would reduce the prevalence of victimization; and (2) building resilience in victims so that the negative impact of victimization on their mental health will be reduced. The secondary objective will be to evaluate the moderating role of gender and the degree of development in the effects of the intervention.The study will involve the evaluation of the intervention in a sample of around 600 adolescents randomly allocated to experimental and control condition.

ELIGIBILITY:
Inclusion Criteria:

* Spanish or Basque understanding
* Permission by parents
* Voluntarity

Exclusion Criteria:

-

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 850 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline scores of the Cyber Bullying Questionnaire (CBQ; Calvete et al., 2010; Gámez-Guadix, Villa-George, & Calvete, 2014) | Baseline, 3 months, and 6 months.
  Self reported levels of perpetration (9 items) and victimization (9 items) of peer cyber aggression. Each item is scored 0-4 (0 = never; 4 = almost every week).
Change from baseline scores of the Functional Assessment of Self-Mutilation (FASM; Lloyd, Kelley & Hope, 1997) | Baseline, 3 months, and 6 months.
  Self reported levels of Non-Suicidal Self-Harm (NSSH). The 6 most representative items will be used. Each item is scored 0-4 (0 = 0 times; 4 = > 11 times).
Change from baseline scores of the reduced version of the Center for Epidemiological Studies Depression (CES-D; Rueda-Jaimes et al., 2009). | Baseline, 3 months, and 6 months.
  Self reported symptoms of depression through 10 items, with a four-point response scale ranging from 0 (practically never) to 3 (almost all the time).
Change from baseline scores of the reduced Spanish version of the Social Anxiety Scale for Adolescents (SAS-A; La Greca & Lopez, 1998; Nelemans et al., 2019) | Baseline, 3 months, and 6 months.
  Self reported symptomatology of social anxiety through 12 items, with a five-point response scale ranging from 1 (not at all) to 5 (all the time).
Change from baseline scores of the reduced version of the Eating Attitudes Test (EAT; Garner & Garfinkel, 1979; EAT-8, Richter, Strauss, Braehler, Altmann & Berger, 2016) | Baseline, 3 months, and 6 months.
  Self reported symptomatology associated with eating disorders through 8 items, with a six-point response scale ranging from 1 (never) to 6 (always).

SECONDARY OUTCOMES:
Change from baseline scores of Entity and incremental theories (Levy, Stroessner, & Dweck, 1998). | Baseline, 1 hour, 3 months, and 6 months.
  Entity and incremental theories will be evaluated using eight items adapted to the situations of bullying in schools. Items are rated on a six-point scale ranging from 1 (strongly disagree) to 6 (strongly agree).
Change from baseline scores of attitude towards cyberbullying measure | Baseline, 1 hour, 3 months, and 6 months.
  Self reported ad hoc measures developed by the research team of the attitude towards cyberbullying. The participants will classify one situation of cyberbullying through adjectives using the semantic differential technique with a response range of 7 points.
Change from baseline scores of attitude towards different courses of action measure | Baseline, 1 hour, 3 months, and 6 months.
  Self reported ad hoc measures developed by the research team of the attitude towards different courses of action when the adolescent witnesses cyberbullying. The participants will rate four different ways to react to cyberbullying through semantic differential items.
Change from baseline scores of the anticipation of reactions and behaviors measure | Baseline, 1 hour, 3 months, and 6 months.
  Self reported ad hoc measures developed by the research team of the anticipation of reactions and behaviors when the adolescent is a witness. The participants will answer seven items on a five-point response scale ranging from 0 (totally disagree) to 3 (totally agree).
Change from baseline scores of the intention to use different strategies when the adolescent is exposed to diverse stressors | Baseline, 1 hour, 3 months, and 6 months.
  Self reported ad hoc measures developed by the research team of the intention to use different strategies when the adolescent is exposed to diverse stressors, participants will complete six items on a four-point response scale ranging from 0 (never or almost never) to 3 (always or almost always).

CONTACTS AND LOCATIONS:
Overall Officials: Esther Calvete, PhD, Principal Investigator — University of Deusto
Locations (1):
- University of Deusto, Bilbao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be available at OSF when the results of the study are published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol and informed consent protocol will be published at clinicaltrials.org Data will be available at OSF when the results are published.
Access Criteria: Public

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-31): https://cdn.clinicaltrials.gov/large-docs/31/NCT04509531/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-31): https://cdn.clinicaltrials.gov/large-docs/31/NCT04509531/ICF_001.pdf